CLINICAL TRIAL: NCT04291898
Title: Comparative Effectiveness of Three Devices for Transcatheter Closure of Atrial Septal Defects for Adults: A Pilot Study (Trio-ASD)
Brief Title: Comparison of Devices for Atrial Septal Defects Closure: A Pilot Study
Acronym: Trio-ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Montreal Heart Institute (Other); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other); St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Eric Horlick, Interventional and Congenital Cardiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-6095; TrioASD (Other: UHN)
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Atrial Septal Defect
Keywords: Transcatheter; Closure; Percutaneous; Atrial Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of three arms for the duration of the study. The arms include: ASO, FSO, GAO/GSO which indicate the type of intervention they will be receiving.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients and outcome assessors will be blinded to the device they receive. Healthcare providers or site coordinators cannot be blinded due to clear differences between devices.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Device: ASO (Active Comparator): Participants implanted with the AMPLATZER™ Septal Occluder (ASO)
  Interventions: Device: AMPLATZER™ Septal Occluder.
- Device: FSO (Active Comparator): Participants implanted with the Occlutech Figulla Flex II® (FSO).
  Interventions: Device: Occlutech Figulla Flex II®
- Device: GSO/GAO (Active Comparator): Participants implanted with the GORE® CARDIOFORM ASD Occluder (GSO/GAO)
  Interventions: Device: GORE® CARDIOFORM ASD Occluder

INTERVENTIONS:
Device: AMPLATZER™ Septal Occluder. — Implantation of the AMPLATZER™ Septal Occluder in the ASD.
  Arms: Device: ASO
Device: Occlutech Figulla Flex II® — Implantation of the Occlutech Figulla Flex II® in the ASD.
  Arms: Device: FSO
Device: GORE® CARDIOFORM ASD Occluder — Implantation of the GORE® CARDIOFORM ASD Occluder or GORE® CARDIOFORM Septal Occluder in the ASD.
  Arms: Device: GSO/GAO

SUMMARY:
This is a proposal, for the first time in Canada, to examine the comparative effectiveness of three commercially available devices (ASO, FSO, and GAO/GSO) for transcatheter closure of atrial septal defects (ASD) in adults using a pilot randomized controlled trial.

DETAILED DESCRIPTION:
The most widely used transcatheter device for ASD closure is the the Amplatzer Septal Occluder (ASO). Two other devices that entered the Canadian market are the Gore Cardioform ASD occluder (GAO) and the Figulla Flexible II Occlutech (FSO) device. There exists a paucity of data on the comparative efficacy and safety of these devices. This is a proposal, for the first time in Canada, to examine the comparative effectiveness of three commercially available ASD devices in an internal pilot randomized trial.

Approximately 60 patients referred for transcatheter ASD closure will be recruited in this study over a period of 15 months from 4 participating centers across Canada. This will be a registry-based randomized controlled trial (RRCT) where patients will be enrolled into one of three arms (ASO, FSO, and GAO/GSO) to compare the effectiveness and safety outcomes of three different ASD closure devices.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old referred for percutaneous (secundum) ASD closure with right atrial and ventricular enlargement; and
* clinically significant left-to-tight shunt (Qp:Qs≥1.5:1), or
* evidence of paradoxical embolism (with a TEE defect >10mm),
* written informed consent

Exclusion Criteria:

* TEE/CCT/CMR defect diameter >30mm,
* rim sizes of < 5 mm to the coronary sinus, inferior vena cava rim, an atrioventricular valve, or the right upper pulmonary vein,
* multiple defects,
* complex congenital heart disease requiring surgical repair within 3 years of device placement,
* Eisenmenger-syndrome,
* recent myocardial infarction PCI/CABG < 6 weeks,
* demonstrated intra cardiac thrombi on echocardiography (especially LA or LAA thrombi), or atrial tumor
* known occluded bilateral femoral veins/IVC,
* pulmonary artery systolic pressure more than half the systemic systolic arterial pressure
* recent pelvic venous thrombosis
* serious comorbidity with life expectancy <3 years (e.g., non-skin cancers not in remission, advanced renal failure serum creatinine >160 umol/L)
* patients whose size or condition would cause the patient to be a poor candidate choice for cardiac catheterization (e.g., too small for echocardiographic imaging probe, catheter size, vascular size, active infection, body weight < 8 kg)
* serious infection in < 6 weeks producing bacteremia (e.g. sepsis), active endocarditis, or any other infection that cannot be treated successfully prior to device implantation (patient must have negative blood cultures off antibiotics for 1 week prior to procedure),
* active GI bleed < 6 weeks,
* bleeding disorder, untreated ulcer, or any other contraindications to aspirin therapy, unless another antiplatelet agent can be administered for 6 months
* previous stroke in the past 12 months,
* documented chronic atrial fibrillation or >2 episodes of documented paroxysmal atrial fibrillation in the last 12 months,
* pregnancy or breastfeeding, plan to become pregnant within the next 6 months, not using an effective method of birth control in premenopausal women,
* documented nickel/titanium allergy, or intolerance to contrast agents.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of 'Clinical atrial fibrillation (AF)' or 'Major adverse cerebro-cardiovascular events (MACCE) | 24 weeks
  At 24 weeks where clinical (AF) includes AF-related, ECG-documented, ED visit/hospitalization/physician visit, cardioversion, ablation or pacemaker implantation or new antiarrhythmic or AF anticoagulant prescription'; MACCE includes 'new onset heart failure (HF), HF-related ED admission, myocardial infarction, stroke, re-intervention, or death.

SECONDARY OUTCOMES:
Subclinical AF (SCAF) burden (days): | 14 days
  Days with >6 min of AF detected on CardioSTAT monitor during 14 days
Subclinical AF (SCAF) burden (number of episodes): | 14 days
  Number of episodes with >6 min of AF detected on CardioSTAT monitor during 14 days
Subclinical AF (SCAF) burden (total time): | 14 days
  Total time in AF during 14 days
Subclinical AF (SCAF) burden (percent time): | 14 days
  Percent time in AF during 14 days
Procedural effectiveness outcomes (acute technical success rate at discharge) | Discharge, 24 weeks
  Successful deployment and retention without major device related complications, stroke, myocardial infarction (MI) or arrhythmia requiring antiarrhythmic drug or cardioversion
Procedural effectiveness outcomes (successful closure rate at discharge): | Discharge, 24 weeks
  Negative bubble study or residual shunt <2mm
Patient-reported outcomes (QoL): | Baseline, 6 weeks, 24 weeks
  Quality of life (QoL) using the EuroQoL (EQ-5D-5L™) at baseline, 6 weeks, 24 weeks
Patient-reported outcomes (healthcare utilization): | Baseline, 6 weeks, 24 weeks
  Healthcare utilization (ED admission, physician visit, etc) at 6 and 24 weeks
Patient-reported outcomes (SF-12): | Baseline, 6 weeks, 24 weeks
  Quality of life (QoL) using the SF-12 questionnaire at baseline, 6 weeks, 24 weeks
Patient-reported outcomes (HeartQOL): | Baseline, 6 weeks, 24 weeks
  Quality of life (QoL) using the HeartQOL questionnaire at baseline, 6 weeks, 24 weeks
Patient-reported outcomes (satisfaction with device): | 24 weeks
  Satisfaction with the use of CardioSTAT and KardiaMobile devices using a Likert scale at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Horlick, MD, Principal Investigator — University Health Network, Peter Munk Cardiac Centre; Lusine Abrahamyan, MD, PhD, Principal Investigator — University Health Network, Theta Collaborative
Locations (4):
- Canada (4):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montreal (MHI), Montreal, Quebec
  - Institut Universitaire de Cardiologie Et Pneumologie de Quebec/Hopital Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No